CLINICAL TRIAL: NCT04043754
Title: Periodontal Regeneration With Platelet-rich Fibrin (Prf) and Autogenous Bone Graft (Abg) Versus Membrane and Abg in the Treatment of Intrabony Periodontal Defects a Longitudinal Randomized Control Clinical Study
Brief Title: Platelet-rich Fibrin and Autogenous Bone vs Membrane and Autogenous Bone in Intrabony Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Michele Paolantonio, Head of Periodontology, G. d'Annunzio University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 062019
Record Dates: First submitted 2019-07-30; First posted 2019-08-02 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Periodontal Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRF treated patients (Experimental): Periodontal surgery with Platelet Rich Fibrin is performed, after local anaesthesia, mucoperiosteal SPPFs will be raised. Autogenous corticocancellous BG material will be collected using bone scrapers , the PRF membrane cut into small pieces and mixed with the ABG will be placed within the IBDs until they will be completely filled. Then the other two PRF membranes in each patient will be adapted over the grafted defect Finally horizontal mattress and interrupted sutures will be carried out.
  Interventions: Procedure: Periodontal surgery with Platlet Rich fibrin
- GTR treated patients (Active Comparator): Periodontal surgery with MEMBRANE is performed, after local anaesthesia, mucoperiosteal SPPFs will be raised. Autogenous corticocancellous BG material will be collected using bone scrapers ; then, ABG will be applied alternatively with MEMBRANE into the IBD according to the "sandwich" technique until the IBD will be completely filled. Finally the flap will be repositioned and sutures completed by interrupted sutures.
  Interventions: Procedure: Procedure/Surgery: Periodontal surgery with Membrane

INTERVENTIONS:
Procedure: Procedure/Surgery: Periodontal surgery with Membrane — Patients will be treated by periodontal surgical flaps with the addition of Membrane+ bone graft
  Arms: GTR treated patients
Procedure: Periodontal surgery with Platlet Rich fibrin — Patients will be treated by periodontal surgical flaps with the addition of PRF + bone graft
  Arms: PRF treated patients

SUMMARY:
Currently, the most positive documented outcomes of periodontal regenerative therapy (PRT) in intrabony defects (IBDs) have been achieved with a combination of bone grafts ( BGs) and a regeneration material like membranes in guided tissue regeneration ( GTR) technique. Among the graft materials only autogenous bone grafts ( ABGs).and demineralized freeze-dried bone allografts (DFDBA), are considered regenerative materials.

Polypeptide growth factors revealed a potential application in PRT periodontal because are the biological mediators during wound healing and regeneration and autologous platelet concentrates ( PC) constitute a safe and convenient approach to deliver them.

Among PC, platelet-rich fibrin ( PRF) belongs to a group of second-generation blood autologous products prepared by peripheral blood centrifugation without any nonclotting agent, so to obtain a dense three-dimensional clot architecture that concentrates platelets, fibrin, leukocytes, cytokines, and sustain cellular migration. This clot is then compressed to obtain elastic and very strong membranes that can be used directly as membranes or as an agent, after chopping, alone or in combination with BGs.

Several studies demonstrate that PRF is effective in promoting bone regeneration (BR) when used alone or in combination with BG during oral/ periodontal surgery.

To date, there are very few published clinical controlled trials that compare the results of PRF + BGs to the outcomes of PRF / BG alone in the treatment of IBDs and no study about PRF + ABG in the same defects. Only one case report tested the use of PRF + ABG mixed with bovine hydroxyapatite in the treatment of insufficient alveolar ridge width in aesthetic area. The aim of the present study is to verify if the combined use of PRF + ABG in the management of IBDs may be a treatment modality clinically "not inferior" to that with Membrane + ABG.

DETAILED DESCRIPTION:
This is a prospective, randomized and controlled clinical trial designed to evaluate the clinical and radiographic outcomes 12 months after two treatment modalities of IBDs: PRF + ABG into defects in the test subjects( TS); membrane + ABG in the control subjects ( CS). The patients enrolled exhibit unfavourable IBDs and all experimental sites will be accessed with a simplified papilla preservation flap ( SPPF) procedure. The filling material (ABG) is common to both treatments: therefore, the investigation will focus on the addictive effect of PRF used in place of MEMBRANE. MEMBRANE is chosen as the active control ( AC) as it is currently considered as the biological "gold standard" agent for the treatment of IBDs.

A non-inferiority trial ( NIT) is designed to prove that using PRF instead of MEMBRANE could achieve a similar result, reducing the treatment's cost and allowing the clinicians to use autogenous material only.

An AC (comparator) is present, but the investigators do not include a third experimental arm, a group of IBDs treated using Open Flap Debridement ( OFD) alone, as it is widely accepted in NITs.

The estimate of the AC effect vs. placebo is assumed from a recent meta-analysis, by the Lower Bound of a 95% Confidence Interval ( CI) of the mean of MEMBRANE + ABG, while an OFD estimate from the corresponding 95%.. The difference between estimates is set as the added benefit of the AC and as a ground for the assay sensitivity.

44 patients affected by moderate-to-severe chronic periodontitis, will be selected for the study. Each patient will participate in the study with a single experimental site. The participants will receive verbal and written information and they will sign a consent form approved by the Ethical Committee of the G. DAnnunzio University of Chieti - medical faculty. The study protocol is in accordance with the Declaration of Helsinki of 1975, revised in Tokyo in 2004. Four months before the surgical treatment, all 44 patients will undergo SRP by ultrasonic instruments and hand curettes and motivational instructions on oral home care.

Non-inferiority margin. A reliable estimate of the expected clinical attachment level ( CAL) gain from an MEMBRANE+ ABG treatment is drawn from a recent meta-analysis, reporting on 548 IBDs in 434 patients.

By literature, CAL gain obtainable by OFD surgical treatments alone is 2.47 mm. The differential effect of using MEMBRANE amounts about 1 .

Each defect will be assigned a defect number and will be randomly allocated to one of the two treatment regimens. Assignment will be performed by a custom made computer-generated table. To conceal allocation, opaque envelopes will be assigned to the specific experimental site and will be opened during surgery Preoperative and 3- 6- 12-months postoperative intraoral standardized radiographs will be taken by the paralleling technique using an individual film-holder device consisting of a bite block rigidly connected to an acrylic dental splint to achieve identical film placement at each evaluation. Pre- and postoperative radiographs will be evaluated by two experienced clinicians who will be masked with respect to the provenience of the radiographs and the clinical measurements. The positions of alveolar crest level and of the bottom of the defect distance and will be marked by a pencil on the radiographs and bottom of the defect will be measured by a millimeter grid. Linear distances between the most coronal interproximal alveolar crest level and the bottom of the defect will be obtained by counting the walls

ELIGIBILITY:
Inclusion Criteria:

* a full-mouth plaque score (FMPS) 25 and a full-mouth bleeding score (FMBS) 26 < 20% at the time of surgery
* to have at least 20 teeth,; at least 1 tooth exhibiting vertical bone loss detected by radiographic examination (alveolar crest level (ACL) - bottom of the defect (BD) distance - -Bone defect depth (BDD) ≥ 4 mm and a probing pocket depth (PPD) ≥ 5mm when evaluated 12 weeks after phase I non- surgical therapy [ scaling and root planing ( SRP)]

Exclusion Criteria:

* no systemic diseases
* no medications affecting periodontal status during the previous 6 months
* not pregnant or lactating; non-smoker
* no periodontal therapy in the 2 previous years, no inadequate endodontic treatment, no dental mobility

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2018-06-10 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Periodontal attachment gain | 6 months
  Change of the distance between the cementum-enamel junction and the depth of the probable site

CONTACTS AND LOCATIONS:
Overall Officials: michele paolantonio, Principal Investigator — università G. D'annunzio Chieti-Pescara
Locations (1):
- G. d'Annunzio University, Chieti, CH, Italy

IPD SHARING:
Plan to Share IPD: No